CLINICAL TRIAL: NCT01111565
Title: A Multicenter, Randomized, Double-blind Study to Evaluate the Efficacy, Safety and Tolerability of an Oral Aripiprazole/Escitalopram Combination Therapy in Patients With Major Depressive Disorder
Brief Title: Study to Evaluate the Efficacy, Safety and Tolerability of an Oral Aripiprazole/Escitalopram Combination Therapy in Participants With Major Depressive Disorder (MDD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated early due to Sponsor decision, closure of this combination therapy program is unrelated to any safety issues, no signals of concern.
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 31-08-263; 2010-018859-97 (EudraCT Number)
Record Dates: First submitted 2010-04-22; First posted 2010-04-27 (Estimated); Results first posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Major Depressive Disorder; MDD; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram; Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase B: Single-blind Prospective Treatment Phase (Experimental): Escitalopram 10 mg capsule, orally, once daily increased to 20 mg/day at the Week 1 (end of Week 1) based upon tolerability profile, for 8 weeks. No dose reductions were allowed after Week 4 and no dose increments were allowed after Week 3. Participants with incomplete response at the end of the Phase B (Week 8) entered Phase C and the rest of the participants continued to Phase B+.
  Interventions: Drug: Escitalopram
- Phase B+: Single-blind Phase B Responders (Experimental): Participants with response (≥50% reduction in depressive symptom severity in HAM-D17 Total Score; or a HAM-D17 Total Score of <14 at Week 8 or a Clinical Global Impression of Improvement (CGI-I) Score of <3 at the Week 6 or 8) at the end of the Phase B (Week 8) continued treatment with the single-blind escitalopram monotherapy at the dose (10 or 20 mg/day) taken during the final week of Phase B, for an additional 6 weeks (Up to Week 14), in Phase B+.
  Interventions: Drug: Escitalopram
- Phase C: Aripiprazole/Escitalopram Combination (Experimental): Participants with incomplete response at Week 8 who were randomized to this arm group received aripiprazole 3, 6, or 12 mg capsule, orally, once daily in combination with the escitalopram 10 or 20 mg orally for 6 weeks (Up to Week 14), in Phase C. No dose adjustments were allowed for escitalopram during Phase C. Participants were titrated to the aripiprazole target dose of 12 mg/day at Week 9 if the initial 6 mg/day dose was tolerated.
  Interventions: Drug: Escitalopram; Drug: Aripiprazole
- Phase C: Escitalopram Monotherapy (Experimental): Participants with incomplete response at Week 8 who were randomized to this arm group received escitalopram monotherapy 10 or 20 mg capsule, orally, once daily, whichever dose was taken during the final week of Phase B for 6 weeks (Up to Week 14), in Phase C. No dose adjustments were allowed for escitalopram monotherapy during Phase C.
  Interventions: Drug: Escitalopram
- Phase C: Aripiprazole Monotherapy (Experimental): Participants with incomplete response at Week 8 who were randomized to this arm group received aripiprazole 3, 6, or 12 mg capsule, orally, once daily for 6 weeks (Up to Week 14), in Phase C. Participants were titrated to the aripiprazole target dose of 12 mg/day at Week 9 if the initial 6 mg/day dose was tolerated. No dose increments were allowed after Week 12; however, doses may have been decreased at any visit, based upon tolerability.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Escitalopram — Escitalopram capsule administered orally, once daily without regard to meals.
  Arms: Phase B+: Single-blind Phase B Responders; Phase B: Single-blind Prospective Treatment Phase; Phase C: Aripiprazole/Escitalopram Combination; Phase C: Escitalopram Monotherapy
Drug: Aripiprazole — Aripiprazole capsule administered orally, once daily without regard to meals.
  Arms: Phase C: Aripiprazole Monotherapy; Phase C: Aripiprazole/Escitalopram Combination

SUMMARY:
This will be a multicenter, randomized, double-blind study designed to assess the efficacy, safety and tolerability of an oral Aripiprazole/Escitalopram combination therapy in participants with MDD who have demonstrated an incomplete response to a prospective trial of Escitalopram, and report a treatment history for the current MDD episode of an inadequate response to at least one and no more than three adequate trials of an approved antidepressant other than Escitalopram. An inadequate response is defined as less than a 50% reduction in depressive symptom severity as assessed by the participant's self-report on the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (ATRQ) and evaluated by the investigator as part of the participant's medical and psychiatric history. An adequate trial is defined as an antidepressant treatment for at least 6 weeks duration (or at least 3 weeks for combination treatments) at an approved dose as specified in the ATRQ.

DETAILED DESCRIPTION:
The study will be organized as follows:

* Screening Phase
* Single-blind Prospective Treatment Phase
* Single-blind Continuation Phase (Responder)or Double-blind Randomization Phase (non-Responder)
* 30 day Post Treatment Follow-up

Assigned Interventions:

* Escitalopram monotherapy
* Aripiprazole/Escitalopram combination therapy
* Aripiprazole monotherapy

ELIGIBILITY:
Inclusion Criteria:

* Participants with a current diagnosis of a major depressive episode. The current depressive episode must be ≥8 weeks in duration
* Participants willing to discontinue all prohibited psychotropic medication starting from the time of signing the informed consent and during the study period
* Participants with a 17-item Hamilton Depression Rating Scale (HAM-D17) Total Score ≥18 at the Baseline for the Prospective Treatment Phase

Exclusion Criteria:

* Lack of prior treatment with an antidepressant during the current depressive episode
* Participants who report treatment with adjunctive or monotherapy antipsychotic treatment during the current depressive episode.
* Participants experiencing hallucinations, delusions or any psychotic symptomatology in the current depressive episode
* Participants with epilepsy or significant history of seizure disorders
* Participants with a clinically significant current diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal or histrionic personality disorder
* Participants who have received electroconvulsive therapy (ECT) in the last 10 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2010-10-04 (Actual); Primary Completion 2011-09-01 (Actual); Study Completion 2011-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (47):
- United States (15):
  - Tucson, Arizona
  - Chino, California
  - Riverside, California
  - Torrance, California
  - Hamden, Connecticut
  - Marietta, Georgia
  - Belmont, Massachusetts
  - Weymouth, Massachusetts
  - Saint Charles, Missouri
  - St Louis, Missouri
  - Brooklyn, New York
  - Garfield Heights, Ohio
  - Philadelphia, Pennsylvania
  - East Providence, Rhode Island
  - Kirkland, Washington
- Canada (3):
  - Penticton, British Columbia
  - Vancouver, British Columbia
  - Burlington, Ontario
- Croatia (3):
  - Osijek
  - Rijeka
  - Zagreb
- France (2):
  - Douai
  - Élancourt
- Hungary (4):
  - Baja
  - Balassagyarmat
  - Budapest
  - Gyula
- India (3):
  - Hyderabad, Andhra Pradesh
  - Visakhapatnam, Andhra Pradesh
  - Mumbai, Maharashtra
- Malaysia (3):
  - Tampoi, Johor Bahru
  - Kajang, Selangor
  - Kuala Lumpur
- Poland (6):
  - Bełchatów
  - Bialystok
  - Study Site 1, Choroszcz
  - Study Site 2, Choroszcz
  - Sosnowiec
  - Tuszyn
- South Africa (4):
  - Study Site 1, Cape Town
  - Study Site 2, Cape Town
  - Durban
  - Pretoria
- Spain (2):
  - Barcelona
  - Salamanca
- Sweden (2):
  - Gothenburg
  - Malmo

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 70 investigative sites in the United States, Canada, France, India, Malaysia, Poland, and South Africa from 4 October 2010 to 1 September 2011.
Pre-assignment Details: A total of 137 participants were enrolled in Phase B (Single-blind Prospective Treatment Phase) to receive escitalopram monotherapy(10 or 20mg/day),of which 26 responders continued to Phase B+(Single-blind Phase B Responders),received escitalopram monotherapy(10 or 20mg/day).45 non-responders were randomized in 1:1:1 ratio to Phase C(Double-blind Randomization Phase),received aripiprazole/escitalopram combination therapy or escitalopram or aripiprazole monotherapy.
Period: Phase B (Weeks 0 to 8)
Arm/Group | Phase B: Single-blind Prospective Treatment Phase | Phase B+: Single-blind Phase B Responders | Phase C: Aripiprazole/Escitalopram Combination | Phase C: Escitalopram Monotherapy | Phase C: Aripiprazole Monotherapy
Started | 137 | 0 | 0 | 0 | 0
Completed | 71 | 0 | 0 | 0 | 0
Not Completed | 66 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Sponsor Discontinued Study | 58 | 0 | 0 | 0 | 0
Not completed — Investigator Withdrew Subject | 1 | 0 | 0 | 0 | 0
Not completed — Subject Withdrew Consent | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy as Determined by the Investigator | 1 | 0 | 0 | 0 | 0
Period: Phase B + and Phase C (Weeks 9 to 14)
Arm/Group | Phase B: Single-blind Prospective Treatment Phase | Phase B+: Single-blind Phase B Responders | Phase C: Aripiprazole/Escitalopram Combination | Phase C: Escitalopram Monotherapy | Phase C: Aripiprazole Monotherapy
Started | 0 | 26 | 16 | 14 | 15
Completed | 0 | 19 | 11 | 10 | 11
Not Completed | 0 | 7 | 5 | 4 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0
Not completed — Sponsor Discontinued Study | 0 | 7 | 3 | 2 | 3
Not completed — Investigator Withdrew Subjects | 0 | 0 | 0 | 1 | 0
Not completed — Subjects Withdrew Consent | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Phase B Sample included all participants who took at least one dose of escitalopram as indicated on the dosing record.
Arm/Group | Phase B: Single-blind Prospective Treatment Phase
Number analyzed (Participants) | 137
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 129
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 26
  White | 90
  More than one race | 0
  Unknown or Not Reported | 11

OUTCOME MEASURES:

1. Primary Outcome: Phase C: Mean Change From End of Phase B (Week 8) in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score to End of Phase C (Week 14)
Description: The MADRS assessed severity of depressive symptoms. It ranges from a minimum of 0 to a maximum of 60 (higher scores indicating a greater severity of depressive symptoms). Participants are rated on 10 items (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and a lack of interest) each on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). A negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms. Last observation carried forward (LOCF) method was used for analyses.
Time Frame: Week 8 to Week 14
Population: Intent-to-treat (ITT) Sample included all participants in the Randomized Sample who received at least one dose of double blind trial medication and had at least one post-randomization efficacy evaluation in Phase C.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase C: Aripiprazole/Escitalopram Combination | Phase C: Escitalopram Monotherapy | Phase C: Aripiprazole Monotherapy
Number analyzed (Participants) | 16 | 14 | 15
score on a scale | -9.0 (2.1) | -3.6 (2.2) | -3.8 (2.1)
Statistical Analysis 1: Comparison: Phase C: Aripiprazole/Escitalopram Combination vs Phase C: Escitalopram Monotherapy; Test type: Superiority; p = 0.079, ANCOVA; Treatment Difference = -5.4, 95% CI 2-sided [-11.5 to 0.7]
Statistical Analysis 2: Comparison: Phase C: Aripiprazole/Escitalopram Combination vs Phase C: Aripiprazole Monotherapy; Test type: Superiority; p = 0.085, ANCOVA; Treatment Difference = -5.2, 95% CI 2-sided [-11.2 to 0.7]

2. Secondary Outcome: Phase C: Clinical Global Impression - Improvement Scale (CGI-I) Score at the End of Phase C
Description: CGI-I is a 7-point clinician-rated scale ranging from 1 to 7, rated as 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. A higher score indicates greater impairment. LOCF method was used for analyses.
Time Frame: Week 14
Population: ITT Sample included all participants in the Randomized Sample who received at least one dose of double blind trial medication and had at least one post-randomization efficacy evaluation in Phase C.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Phase C: Aripiprazole/Escitalopram Combination | Phase C: Escitalopram Monotherapy | Phase C: Aripiprazole Monotherapy
Number analyzed (Participants) | 16 | 14 | 15
score on a scale | 2.5 (0.2) | 3.0 (0.2) | 2.9 (0.2)
Statistical Analysis 1: Comparison: Phase C: Aripiprazole/Escitalopram Combination vs Phase C: Escitalopram Monotherapy; Test type: Superiority; p = 0.148, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel Row Mean Scores Test was used to determine the p-value; Treatment Difference = -0.5, 95% CI 2-sided [-1.1 to 0.1]
Statistical Analysis 2: Comparison: Phase C: Aripiprazole/Escitalopram Combination vs Phase C: Aripiprazole Monotherapy; Test type: Superiority; p = 0.242, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel Row Mean Scores Test was used to determine the p-value; Treatment Difference = -0.4, 95% CI 2-sided [-1.0 to 0.3]

3. Secondary Outcome: Phase C: Mean Change From End of Phase B (Week 8) in the Sheehan Disability Scale (SDS) Mean Score to End of Phase C (Week 14)
Description: SDS is a 3-item clinician-rated questionnaire used to evaluate impairments in the domains of work, social life/leisure, and family life/home responsibility. The participant is asked to rate the degree to which their functioning is impaired on an 11-point scale, ranging from 0 (not at all) to 10 (extremely). Scores of 0 to 3 indicate mild functional impairment, 4 to 6 indicate moderate functional impairment, and 7 to 9 indicate marked functional impairment. The scores for the 3 domains are summed into a total score that ranges from 0 (unimpaired) to 30 (highly impaired). A higher score indicates greater impairment. A negative change score indicates improvement. LOCF method was used for analyses.
Time Frame: Week 8 to Week 14
Population: ITT Sample included all participants in the Randomized Sample who received at least one dose of double blind trial medication and had at least one post-randomization efficacy evaluation in Phase C. Overall number of participants analyzed are participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase C: Aripiprazole/Escitalopram Combination | Phase C: Escitalopram Monotherapy | Phase C: Aripiprazole Monotherapy
Number analyzed (Participants) | 14 | 13 | 14
score on a scale | -1.6 (0.7) | -1.8 (0.7) | -0.6 (0.7)
Statistical Analysis 1: Comparison: Phase C: Aripiprazole/Escitalopram Combination vs Phase C: Escitalopram Monotherapy; Test type: Superiority; p = 0.910, ANCOVA; Treatment Difference = 0.1, 95% CI 2-sided [-1.8 to 2.1]
Statistical Analysis 2: Comparison: Phase C: Aripiprazole/Escitalopram Combination vs Phase C: Aripiprazole Monotherapy; Test type: Superiority; p = 0.291, ANCOVA; Treatment Difference = -1.0, 95% CI 2-sided [-3.0 to 0.9]

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 30 days after the last dose of study drug (up to approximately 22 weeks)
Description: Phase B Sample included all participants who took at least one dose of escitalopram as indicated on the dosing record. Phase B+ Sample included all participants who responded at the end of Phase B (were therefore not randomized) and who continued on single-blind escitalopram beyond Week 8. Randomized Sample included all participants who were randomized in Phase C.
Arm/Group | Phase B: Single-blind Prospective Treatment Phase | Phase B+: Single-blind Phase B Responders | Phase C: Aripiprazole/Escitalopram Combination | Phase C: Escitalopram Monotherapy | Phase C: Aripiprazole Monotherapy
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/26 | 0/16 | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/137 | 0/26 | 0/16 | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 65/137 | 4/26 | 12/16 | 11/14 | 13/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase B: Single-blind Prospective Treatment Phase (N=137) | Phase B+: Single-blind Phase B Responders (N=26) | Phase C: Aripiprazole/Escitalopram Combination (N=16) | Phase C: Escitalopram Monotherapy (N=14) | Phase C: Aripiprazole Monotherapy (N=15)
Dry mouth (Gastrointestinal disorders) | 7 | 1 | 1 | 1 | 3
Nausea (Gastrointestinal disorders) | 18 | 2 | 2 | 0 | 2
Asthenia (General disorders) | 1 | 0 | 2 | 0 | 1
Fatigue (General disorders) | 7 | 0 | 1 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 3 | 0 | 0
Akathisia (Nervous system disorders) | 1 | 0 | 2 | 1 | 1
Dizziness (Nervous system disorders) | 9 | 0 | 2 | 1 | 1
Headache (Nervous system disorders) | 15 | 0 | 1 | 1 | 2
Lethargy (Nervous system disorders) | 2 | 0 | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 1 | 1 | 2
Restlessness (Psychiatric disorders) | 2 | 0 | 2 | 0 | 4
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Irritability (General disorders) | 2 | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 2 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Drooling (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Sedation (Nervous system disorders) | 2 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 8 | 1 | 1 | 1 | 3
Tremor (Nervous system disorders) | 3 | 0 | 2 | 1 | 0
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Libido decreased (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Middle insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Yawning (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early due to Sponsor decision, closure of this combination therapy program is unrelated to any safety issues, no signals of concern.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.